CLINICAL TRIAL: NCT04080726
Title: A Multicenter, Randomized, Double-blind, Phase Ⅲ Study to Compare Efficacy and Safety of HIP1601 40mg and HGP1705 40mg in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Efficacy and Safety of HIP1601 Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ESOM-301
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Erosive Gastroesophageal Reflux Disease
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-blind, parallel group study
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIP1601+HGP1705 Placebo (Experimental): HIP1601+HGP1705 Placebo for 4weeks. if not fully cured, take HIP1601+HGP1705 Placebo for addtional 4weeks
  Interventions: Drug: HIP1601; Drug: HGP1705 Placebo
- HGP1705+HIP1601 Placebo (Experimental): HGP1705+HIP1601 Placebo for 4weeks. if not fully cured, take HGP1705+HIP1601 Placebo for addtional 4weeks
  Interventions: Drug: HGP1705; Drug: HIP1601 Placebo

INTERVENTIONS:
Drug: HIP1601 — Oral esomeprazole
  Other Names: esomeprazole
  Arms: HIP1601+HGP1705 Placebo
Drug: HGP1705 — Oral Nexium Tab
  Other Names: Nexium Tab
  Arms: HGP1705+HIP1601 Placebo
Drug: HIP1601 Placebo — Oral Placebo
  Arms: HGP1705+HIP1601 Placebo
Drug: HGP1705 Placebo — Oral Placebo
  Arms: HIP1601+HGP1705 Placebo

SUMMARY:
The purpose of this study is to investigate the safety and clinical efficacy of HIP1601 in patients with erosive gastroesphageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* 19≤ age ≤ 75
* Esophago-Gastro-Duodenoscopy LA classification ≥ grade A
* Patients experienced heartburn or acid regurgitation within 7 days of screening day
* Patients understood the consents and purpose of this trial and signed consent form

Exclusion Criteria:

* Has malignancy in the upper gastrointestinal tract, digestive ulcer, bleeding disorder or signs of gastrointestinal bleeding
* Has a severe liver disorder(at screening day, AST or ALT level exceeds 3 times more than normal upper range)
* Has a clinically significant renal failure(at screening day, MDRD eGFP ≤ 59 mL/min/1.73m2 or Serum creatinine >2.0mg/dL)
* Uncontrolled diabetes mellitus
* Before screening EGD, a patient who has taken H2-receptor antagonist or PPI within 2 weeks
* Before screening EGD, a patient who has taken drugs containing following list within 1 weeks : warfarin, anticholinergics for spasmolytic GI, antineoplastic agents, salicylates(except 100mg a day for prevention of cardiovascular disease), steroids, propulsives, sucralfate, NSAIDs, other antacids(e.g. antacids of prostaglandin analogs, antacids of aluminum/magnesium)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Complete healing rate | at 4 weeks or 8 weeks
  percentage of subjects whose erosion is completely cured

SECONDARY OUTCOMES:
Complete healing rate | at 4 weeks
  percentage of subjects whose erosion is completely cured
Complete resolution rate of each symptom in GERD | at 4,8 weeks
Proportion of heartburn-free days, acid regurgitation-free days | at 1, 2, 4, 8 weeks
Proportion of heartburn-free nights, acid regurgitation-free nights | at 1, 2, 4, 8 weeks
Time to sustained resolution heartburn, acid regurgitation | at 4 weeks or 8 weeks
Time to sustained resolution of nocturnal heartburn, nocturnal acid regurgitation | at 4 weeks or 8 weeks
Total number of use of relief drugs and average usage per day | at 4 weeks or 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hunyong Jung, MD, Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lim H, Park JK, Chung H, Lee SH, Park JM, Park JH, Kim GH, Shin SK, Hong SJ, Lee KJ, Park MI, Jung HK, Kim HS, Sung JK, Jeon SW, Choi SC, Moon JS, Kim N, Park JJ, Hong SH, Kim NY, Jung HY. Efficacy and safety of HIP1601 (dual delayed-release esomeprazole) 40 mg in erosive esophagitis compared to HGP1705 (delayed-release esomeprazole) 40 mg: a multicenter, randomized, double-blind, non-inferiority study. BMC Gastroenterol. 2023 Dec 18;23(1):447. doi: 10.1186/s12876-023-03087-6. PMID 38110901